CLINICAL TRIAL: NCT04105309
Title: Implementation Intentions for Weight Loss and Dietary Change in College Students With Overweight and Obesity
Acronym: ImpInt
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jacqueline Hayes, Graduate Student, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201702063
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Obesity
Keywords: Obesity; College Students; Implementation Intentions
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: three-group parallel randomized-controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Implementation Intention (IMP) (Experimental): Following review of a psychoeducational packet regarding making changes for weight loss, all participants were assigned five dietary goals (e.g. avoiding high-fat foods, eating five servings of fruits and vegetables a day) and a goal to weight daily. Participants in the IMP condition formed an implementation intention for each of the goals at the baseline session. Two examples of implementation intentions were provided for each goal as a model. Participants thought about how they would best be able to achieve the outlined goals in their life on a daily basis (goal-aligned behavior), as well as when, where, and how they would initiate these new behaviors (retrieval cue). Participants then created and wrote down a unique implementation intention for each of the goals using the sentence structure "If/When I _______, then I will ______." No repetitions or combinations of implementation intentions were allowed for standardization across participants.
  Interventions: Behavioral: Implementation Intentions
- Enhanced Implementation Intention (IMP+) (Experimental): Participants completed all tasks of the IMP group and additionally, individuals in the IMP+ condition received fluency training and text message reminders. Fluency training occurred weekly using an online survey tool. On fluency training days, participants received a survey link via email, which consisted of six multiple-choice questions for participant's unique implementation intentions. Participants had to correctly identify their matching goal-aligned behavior among three distractor behaviors as quickly as possible and were given corrective feedback if they chose incorrectly. Text messages containing all six implementation intentions as well as goal reminders that were obtained by asking participants to write down their reasons for wanting to lose weight were sent on four days each week of the intervention (16 days total). At baseline, participants chose how text messages were bundled and when they were sent. Text schedules stayed constant across the study.
  Interventions: Behavioral: Implementation Intentions; Behavioral: Fluency Training; Behavioral: Text Messages
- Goal Intentions (GOL) (Active Comparator): Participants in the GOL condition were assigned the five dietary goals and the daily weighing goal. No additional intervention was given.
  Interventions: Behavioral: Goal Intentions

INTERVENTIONS:
Behavioral: Implementation Intentions — Implementation intentions aid in pre-planning and habitualization of behaviors, as they serve to identify the when, where, and how of behaviors leading to goal attainment. Often taking the form of "If/when situation x arises, then I will do y!", implementation intentions can be conceptualized in two parts, namely, an environmental or internal retrieval cue and a goal-directed behavioral response. Implementation intentions are effective because they 1) create a strong association between a retrieval cue and a goal-aligned behavior, increasing the likelihood that the goal-aligned behavior will be retrieved and utilized when the cue is encountered, and 2) increase attention for and cognitive accessibility of the retrieval cue, increasing opportunities for goal-aligned action .
  Arms: Enhanced Implementation Intention (IMP+); Implementation Intention (IMP)
Behavioral: Fluency Training — Fluency training is a learning strategy that requires an individual to perform a skill or demonstrate knowledge repeatedly for both accuracy and response rate; the goal is to enhance automaticity of the response and promote endurance and retention of skills and knowledge over time and in the face of distractors. Participants completed 1 minute fluency training protocol 4 times throughout the study.
  Arms: Enhanced Implementation Intention (IMP+)
Behavioral: Text Messages — SMS reminders sent to phone of implementation intentions 16 times throughout the study.
  Arms: Enhanced Implementation Intention (IMP+)
Behavioral: Goal Intentions — Intentions to complete a goal that do not specify a plan about how to do so (compared to implementation intentions, that do)
  Arms: Goal Intentions (GOL)

SUMMARY:
One in three college students have overweight or obesity and are in need of brief and simple weight loss interventions that complement their unstructured lifestyles. Implementation intentions, a strategy that connects a goal-aligned behavior to a cue, facilitate goal-attainment for a wide variety of health-behaviors, but have not been tested as a stand-alone treatment for weight loss in students. College students with overweight or obesity (N = 95) were randomized to one of three conditions: an implementation intention group (IMP), an enhanced implementation intention group (IMP+) that included text message reminders and fluency training (i.e., training for speed and accuracy), and a control goal intention group (GOL) for four weeks. Participants completed anthropometric and self-report assessments pre- and post-treatment as well as experience-sampling assessments during the study to assess how implementation intentions contribute more directly to behavior change

DETAILED DESCRIPTION:
Obesity poses a serious public health concern. Thirty-five percent of college students are overweight/obese, putting them at increased risk of overweight and obesity in later adulthood. The study of effective interventions for weight loss has been neglected in this population, and those that have been assessed had high attrition due to time burden. Brief interventions are needed for weight loss in students with obesity to improve current weight status and prevent associated comorbidities in later adulthood.

Self-regulatory behaviors are necessary to achieve weight loss goals, specifically goal-striving behaviors that aid in the planning and execution of goal-aligned actions5. Implementation intentions are a widely-utilized self-regulatory goal striving strategy that function by creating a mental link between a critical environmental or internal retrieval cue and a goal-aligned behavior (e.g. "if I want dessert, then I will eat an apple"). Implementation intentions are effective because they 1) create a strong association between a goal-aligned behavior and a retrieval cue for that behavior, increasing the likelihood that the goal-aligned behavior will be accessed and employed when the cue is encountered, and 2) increase attention for and cognitive accessibility of the retrieval cue, thus increasing opportunities for goal-aligned action. Implementation intentions effectively facilitate health-related goal attainment with regard to diet and weight loss. However, mechanisms underlying implementation intentions may weaken when used in applied, naturalistic settings and when multiple implementation intentions are maintained, due to complexity and difficulty of goal achievement. Enhancements that strengthen implementation intention effects should improve use for clinically-relevant diet change and weight loss in applied interventions.

Strengthening these mechanisms via improved encoding and retrieval should help maintain potency.

Fluency training (i.e., training for speed and accuracy) improves encoding and retention of information14,15 and should strengthen the already present link between the cue and the goal-aligned behavior, facilitating employment of the predetermined behavior, even when competing goals are introduced in applied settings. Additionally, external reminders serve to support memory for and increase accessibility of the multiple cues, allowing for maximal opportunities for the goal-aligned behaviors to be retrieved and utilized. Given high use of mobile devices in college students, text message reminders can serve as external reminders in this population and have been used previously to complement implementation intention use.

Thus, this proposal aims to test the efficacy of an implementation intention intervention alone (IMP) and in combination with fluency training and text message reminders (IMP+) against a goal-intention control (GOL) on weight loss and dietary behaviors. A three-group randomized-controlled intervention paradigm will be employed across four weeks. Ecological momentary assessment (EMA), the repeated testing of participants in real time, will be used to provide a more in-depth snapshot of implementation intention usage and its role as the mechanism of change in the intervention. Work to date examining implementation intentions has been limited to the laboratory or has utilized retrospective self-report, which limit external validity and are susceptible to recall bias. This will be the first study to examine implementation intention use with the externally-valid measurement that EMA provides. Additionally, given literature that supports implementation intention use during periods when goal striving is challenged (e.g. negative mood, etc.), the study will additionally assess their efficacy during disruptive internal and external states. At post-treatment, weight and dietary change will be assessed. Students with overweight/obesity wanting to lose weight, but not currently enrolled in a weight loss program, will be assessed. Specifically, the study will:

Specific Aim 1: Evaluate the effects of IMP and IMP+ on weight (Specific Aim 1a) and diet (Specific Aim 1b). Participants in IMP and IMP+ will lose more weight and show greater diet improvements compared to individuals in GOL. Participants in IMP+ will lose more weight and show greater diet improvements compared to participants in the IMP.

Exploratory Aim: Explore effective use of implementation intentions as the underlying mechanism of treatment outcome and their successful employment when distractions threaten goal attainment.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than or equal to 25
* Interest in losing weight
* Own a mobile Smart phone and willing to receive study text messages and download a mobile application

Exclusion Criteria:

* Currently participating in a formal weight loss program
* Meet diagnostic criteria for an eating disorder as measured by the Eating Disorder Diagnostic Scale

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Body Weight | Measured pre- and post-intervention (4 weeks apart)
  kilograms
Relative Body Weight | Measured pre- and post-intervention (4 weeks apart)
  Body Mass Index, calculated using both height and weight

SECONDARY OUTCOMES:
Kilocalorie Consumption | Measured pre- and post-intervention (4 weeks apart)
  Number of kilocalories consumed per day, collected from the Diet History Questionnaire-II
Diet Quality | Measured pre- and post-intervention (4 weeks apart)
  Measured by the Healthy Eating Index, which ranges from 0-100, calculated using information from the Diet History Questionnaire-II

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benyamini Y, Geron R, Steinberg DM, Medini N, Valinsky L, Endevelt R. A structured intentions and action-planning intervention improves weight loss outcomes in a group weight loss program. Am J Health Promot. 2013 Nov-Dec;28(2):119-27. doi: 10.4278/ajhp.120727-QUAN-365. Epub 2013 Apr 26. PMID 23621700
- [Background] Webb TL, Sheeran P. Mechanisms of implementation intention effects: the role of goal intentions, self-efficacy, and accessibility of plan components. Br J Soc Psychol. 2008 Sep;47(Pt 3):373-95. doi: 10.1348/014466607X267010. Epub 2007 Dec 18. PMID 18096108
- [Background] Hagger MS, Luszczynska A. Implementation intention and action planning interventions in health contexts: state of the research and proposals for the way forward. Appl Psychol Health Well Being. 2014 Mar;6(1):1-47. doi: 10.1111/aphw.12017. Epub 2013 Oct 8. PMID 24591064
- [Background] Luszczynska A, Sobczyk A, Abraham C. Planning to lose weight: randomized controlled trial of an implementation intention prompt to enhance weight reduction among overweight and obese women. Health Psychol. 2007 Jul;26(4):507-12. doi: 10.1037/0278-6133.26.4.507. PMID 17605571